CLINICAL TRIAL: NCT00448734
Title: A Phase 1/2 Study of Picoplatin and Docetaxel (With Prednisone) in Subjects With Chemotherapy-Naive Metastatic Hormone-Refractory Prostate Cancer
Brief Title: A Study of Picoplatin and Docetaxel in Subjects With Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Poniard Pharmaceuticals (Industry)
Responsible Party: Robert Earhart, MD, PhD, Poniard Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0502
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: metastatic; hormone-refractory; prostate cancer; picoplatin; platinum drug; chemotherapy; docetaxel
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — amminedichloro(2-methylpyridine)platinum(II); Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The treatment regimen will be the assigned dose of picoplatin plus docetaxel, 60 mg/m2 or 75 mg/m2, once every three weeks, plus prednisone (or prednisolone, if prednisone is not available), 5 mg orally twice daily beginning on day 1 and continuing daily until therapy is discontinued.
  Docetaxel will be given intravenously over 60 minutes, followed 30 minutes later by picoplatin as a 1-2 hour intravenous infusion.
  Interventions: Drug: Picoplatin
- 2 (Active Comparator): Docetaxel
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: Picoplatin — The treatment regimen will be the assigned dose of picoplatin plus docetaxel, 60 mg/m2 or 75 mg/m2, once every three weeks, plus prednisone (or prednisolone, if prednisone is not available), 5 mg orally twice daily beginning on day 1 and continuing daily until therapy is discontinued.
  Docetaxel will be given intravenously over 60 minutes, followed 30 minutes later by picoplatin as a 1-2 hour intravenous infusion.
  Arms: 1
Drug: docetaxel — The treatment regimen will be the assigned dose of picoplatin plus docetaxel, 60 mg/m2 or 75 mg/m2, once every three weeks, plus prednisone (or prednisolone, if prednisone is not available), 5 mg orally twice daily beginning on day 1 and continuing daily until therapy is discontinued.
  Docetaxel will be given intravenously over 60 minutes, followed 30 minutes later by picoplatin as a 1-2 hour intravenous infusion.
  Arms: 2

SUMMARY:
This study will review the safety of picoplatin, a new type of platinum drug, with docetaxel, a drug commonly used in the treatment of prostate cancer. Patients who are eligible for this study will have had a diagnosis of hormone-refractory prostate cancer that has metastasized to other areas of the body, and have not been previously treated with chemotherapy drugs. Picoplatin will be administered in combination with docetaxel and prednisone to identify the maximum tolerated dose (MTD). Patients will receive IV treatments of picoplatin with docetaxel every 3 weeks, with prednisone, 5 mg orally, twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Radiologic evidence of metastatic disease (Jewett-Whitmore Stages D1-D2 or TNM Stage N1-3 or M1).
* Disease progression or recurrence documented by either: increasing serum PSA on three consecutive measurements each obtained at least one week apart, or findings on radiographic imaging studies.
* Non-surgically castrate subjects must be receiving androgen ablation therapy as maintenance therapy.
* Adequate hormonal therapy as documented by a castrate level of serum testosterone (all subjects without surgical castration must have a serum testosterone less than 50 ng/ml).
* At least 4 weeks must have elapsed after the withdrawal of antiandrogens (6 weeks in the case of bicalutamide).
* Age 18 years and over. Subjects older than 80 years should be entered on study only if considered "physiologically appropriate" for combination chemotherapy.
* ECOG performance score (PS) of 0 or 1.
* Stable levels of pain for at least 7 days before study entry.
* Life expectancy more than 3 months.
* At least 28 days must have elapsed since prior radiotherapy.
* At least 28 days must have elapsed since any prior investigational agent.
* Absolute neutrophil count (ANC) at least 1.5 x 10^9th/L.
* Platelet count at least 100 x 10^9th/L.
* Hemoglobin at least 10 g/dL.
* Serum AST and ALT levels ≥ 1.5 times upper limit of normal (ULN).
* Serum bilirubin ≤ ULN.
* Serum creatinine ≤ ULN.
* All subjects must agree to use appropriate birth control methods while on study and until 1 month after completion of study chemotherapy.

Exclusion Criteria:

* Prior treatment with cytotoxic agents (except estramustine), radioisotopes, or biological therapies other than hormones.
* Clinical evidence of brain or leptomeningeal metastases.
* Symptomatic peripheral neuropathy of Grade 2 or higher.
* History of another cancer within the preceding 5 years, except for superficial skin cancers.
* Known hypersensitivity to drugs formulated with Polysorbate 80.
* Prior radiotherapy that included ≥ 30% of the bone marrow (e.g., the whole of the pelvis or half of the spine).
* Uncontrolled intercurrent illness (e.g., active infection).
* Serious medical or psychiatric illness that could potentially interfere with the completion of the study treatment according to this protocol.
* History of serious cardiac disease, defined as myocardial infarction within six months of enrollment, congestive heart failure classified by the New York Heart Association as Class III or IV, uncontrolled cardiac arrhythmias, poorly controlled or unstable angina, or electrocardiographic evidence of acute ischemia.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
In Part 1, the Maximum Tolerated Dose (MTD) will be determined | MTD
In Part 2, PSA response will be measured (reduction of at least 50% of PSA from baseline, with reduction maintained for at least 4 weeks) | response

SECONDARY OUTCOMES:
Progression free survival | progression

CONTACTS AND LOCATIONS:
Overall Officials: Robert Earhart, MD, Study Director — Poniard Pharmaceuticals
Locations (11):
- Russia (11):
  - Medical Radiology Research Center under the Russian Academy of Medical Sciences, Obninsk, Kaluga Oblast
  - Chelyabinsk Regional Oncology Center, Chelyabinsk
  - Burdenko Central Military Clinical Hospital, Moscow
  - Russian Research Center of Radiology, Moscow
  - Research Institute of Urology - Ministry of Health, Moscow
  - Leningrad Regional Oncology Center, Saint Petersburg
  - Central Medical Unit #122, Saint Petersburg
  - Therapeutic and Research Medical Center, Saint Petersburg
  - St. Petersburg City Hospital #26, Saint Petersburg
  - St. Petersburg City Oncology Center, Saint Petersburg
  - State Medical Institution of Yaroslavl Region / Regional Clinical Oncology Hospital, Yaroslavl

REFERENCES:
- [Background] Beale P, Judson I, O'Donnell A, Trigo J, Rees C, Raynaud F, Turner A, Simmons L, Etterley L. A Phase I clinical and pharmacological study of cis-diamminedichloro(2-methylpyridine) platinum II (AMD473). Br J Cancer. 2003 Apr 7;88(7):1128-34. doi: 10.1038/sj.bjc.6600854. PMID 12671715
- [Background] Canobbio L, Guarneri D, Miglietta L, Decensi A, Oneto F, Boccardo F. Carboplatin in advanced hormone refractory prostatic cancer patients. Eur J Cancer. 1993;29A(15):2094-6. doi: 10.1016/0959-8049(93)90040-m. PMID 7507687
- [Background] Douillard JY, Schiller J. ZD0473 combined with other chemotherapeutic agents for the treatment of solid malignancies. Eur J Cancer. 2002 Dec;38 Suppl 8:S25-31. doi: 10.1016/s0959-8049(02)80020-x. PMID 12645909
- [Background] Gelmon KA, Stewart D, Chi KN, Chia S, Cripps C, Huan S, Janke S, Ayers D, Fry D, Shabbits JA, Walsh W, McIntosh L, Seymour LK. A phase I study of AMD473 and docetaxel given once every 3 weeks in patients with advanced refractory cancer: a National Cancer Institute of Canada-Clinical Trials Group trial, IND 131. Ann Oncol. 2004 Jul;15(7):1115-22. doi: 10.1093/annonc/mdh278. PMID 15205207
- [Background] Holford J, Raynaud F, Murrer BA, Grimaldi K, Hartley JA, Abrams M, Kelland LR. Chemical, biochemical and pharmacological activity of the novel sterically hindered platinum co-ordination complex, cis-[amminedichloro(2-methylpyridine)] platinum(II) (AMD473). Anticancer Drug Des. 1998 Jan;13(1):1-18. PMID 9474239
- [Background] Holford J, Sharp SY, Murrer BA, Abrams M, Kelland LR. In vitro circumvention of cisplatin resistance by the novel sterically hindered platinum complex AMD473. Br J Cancer. 1998;77(3):366-73. doi: 10.1038/bjc.1998.59. PMID 9472630
- [Background] Rogers P, Boxall FE, Allott CP, Stephens TC, Kelland LR. Sequence-dependent synergism between the new generation platinum agent ZD0473 and paclitaxel in cisplatin-sensitive and -resistant human ovarian carcinoma cell lines. Eur J Cancer. 2002 Aug;38(12):1653-60. doi: 10.1016/s0959-8049(02)00107-7. PMID 12142057
- See also: Poniard Pharmaceuticals, Inc. — http://www.poniard.com